CLINICAL TRIAL: NCT06441149
Title: The Impact of a Personalized Data-Based Bronchoscopy Simulation Operation System on Perioperative Anxiety and Satisfaction in Bronchoscopy：a Randomised Controlled Trial
Brief Title: Individualized Data-based High Simulation of Bronchoscopy Operations in Preoperative Bronchoscopy Informed Consent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-AI-informed consent
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Bronchoscopy
Keywords: Communication; Informed Consent; Physician-Patient Relations; AI; bronchoscopy
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard informed consent (Experimental): standard informed consent
  Interventions: Other: Standard informed consent
- AI-based informed consent (Experimental): Patients receiving personalized data-based informed consent procedure before bronchoscopy
  Interventions: Other: AI-based informed consent

INTERVENTIONS:
Other: AI-based informed consent — Patients receiving personalized data-based informed consent procedure before bronchoscopy
  Arms: AI-based informed consent
Other: Standard informed consent — Standard informed consent
  Arms: standard informed consent

SUMMARY:
A prospective randomized controlled study was conducted to investigate whether preoperative replacement of patients based on AI training instruments could alleviate preoperative anxiety.

Patients who met the criteria were randomly assigned to either the personalized data-based group or the control group. Prior to the preoperative account examination, each patient's anxiety level was assessed, after which a 30-40-minute informed consent form was read.

The traditional group underwent a preoperative account and question-and-answer session with an experienced bronchoscopy laboratory physician, after which the scale was reassessed.

The experimental group underwent a simulated surgical procedure on an AI simulation instrument based on the patient's CT personalized data, performed by an experienced bronchoscopist. The bronchoscopist explained the surgical precautions and answered the patient's questions throughout the procedure. Following the responses to the questions, the scale was reassessed. Following surgery, patients are invited to complete a satisfaction survey prior to discharge or following the discussion of bronchoscopy findings.

ELIGIBILITY:
Inclusion Criteria:

* requiring elective bronchoscopy
* Older than 18 years

Exclusion Criteria:

· Dementia, limited speech, or other problems affecting communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
The level of the patient's anxiety | 1 days before Bronchoscopic procedures
  The modified APAIS questionnaire and the VAS scale were employed to assess anxiety levels before and after informed consent.

SECONDARY OUTCOMES:
The level of the patient's satisfication | 1 days after Bronchoscopic procedures
  The post-surgical satisfaction questionnaire consisted of four questions on a 5-point Likert scale, with responses ranging from "strongly agree" to "strongly disagree."

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China